CLINICAL TRIAL: NCT01753817
Title: Observational Study of Radial Artery Patency Following Catheterization With a 7F Sheath
Brief Title: Assessment of Radial Artery Patency Following Catheterization With a 7F Sheath
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jaffe, Ronen, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: CMC-12-0016 CTIL
Record Dates: First submitted 2012-12-18; First posted 2012-12-20 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Catheterization; Transradial Patency
Keywords: Coronary catheterization; Transradial patency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort: Cohort of patients who have previously undergone transradial catheterization with the use of a 7F vascular sheath

SUMMARY:
Radial artery occlusion may occur after performance of coronary catheterization via the radial artery (transradial approach). In some cases it may be desirable to insert large (7F) catheters via the radial artery, however the impact of increased catheter size on subsequent radial artery patency is unclear. We hypothesize that radial artery occlusion following 7F catheterization is rare and occurs in < 5% of the cases.

DETAILED DESCRIPTION:
Background:

Coronary catheterization is a commonly performed diagnostic and therapeutic procedure. The procedure is most commonly performed via the transfemoral approach (via the femoral artery). Recently the transradial approach (via the radial artery) has been gaining popularity since it is associated with decreased risk of bleeding and facilitates patient mobilization following the procedure (1-3). During the catheterization procedure a sheath (tube) is inserted into the access artery so as to enable insertion of catheters and devices into the body. Vascular sheaths may have different internal diameters, which are measured in French (F) units. Commonly used sheath sizes for coronary catheterization are 5F and 6F, however use of larger 7F sheaths is beneficial when more complex procedures are performed such as insertion of two coronary stents. Use of a 7F sheath creates a slightly larger orifice within the blood vessel wall and may potentially increase the risk of damage to the vessel wall and hemorrhage.

The palm of the hand normally receives dual blood supply via the radial and ulnar arteries. Prior to performing transradial catheterization the ability of the ulnar artery to supply blood to the whole palm is confirmed by performing an Allen Test, in order to avoid palmar ischemia if the radial artery becomes occluded following the procedure. Radial artery occlusion in the presence of a normal pre-procedural Allen Test is almost universally asymptomatic, however it may preclude future use of the radial artery for vascular access or as a coronary graft if bypass surgery is performed. The frequency of radial artery occlusion following transradial catheterization ranges from 5% to 15% in different reports (4), depending on many factors such patient selection, degree of anticoagulation during the procedure and the time interval between performance of the procedure and studying the radial artery patency. Use of larger sheaths has also been reported as a risk factor for radial artery occlusion (5), however the true incidence of this complication is unclear. It is desirable to discover the true rate of radial artery occlusion following catheterization with a 7F sheath, since such knowledge may assist physicians in planning the optimal catheterization strategy.

Aims:

The aim of the study will be to examine the occurrence of radial artery occlusion following transradial catheterization with a 7F sheath.

Hypothesis:

Radial artery occlusion following 7F catheterization is rare and occurs in < 5% of the cases.

Methods:

The study will be performed as part of Mr. Dan Levin's required Medical School Thesis research at the Faculty of Medicine, Technion IIT, Haifa, Israel. Two-hundred subjects who have previously undergone transradial catheterization between the years 1999 and 2012 with a 7F sheath will be identified in the Lady Davis Carmel Medical Center Catheterization laboratory computerized database. The subjects will be contacted by the study investigators and will be invited to a meeting with the investigators at Carmel Medical Center. The study protocol consists of a single meeting between the investigators and the study subjects. During this meeting the subjects will be given explanation of the study protocol. If they consent to participate in the study they will sign an informed consent form, undergo physical examination of the reverse Allen test and ultrasound examination of the patency of the radial artery. Radial artery patency will be studied with the reverse Allen test. This test is performed by simultaneously occluding both the radial and ulnar arteries until no pulse signal is detected with a pulse oximeter placed on the index finger. The pressure on the radial artery is then released and reappearance of the pulse signal on the oximeter is documented-signifying antegrade flow in the radial artery. This test is not associated with any reported complications or morbidity. Radial artery flow will be studied with Doppler ultrasound. The ultrasound test will be performed by Dr Salim Adawi at no cost. The ultrasound test is a routine non-invasive study which is not associated with any reported complications or morbidity. Clinical and procedural data will be collected in the CRF form in order to characterize risk factors for radial artery occlusion.

Endpoints:

1. Normal reverse Allen test.
2. Antegrade flow in the radial artery by ultrasound.

Number of participants:

The Lady Davis Carmel Medical Center catheterization laboratory database will be scanned in order to identify all patients who have undergone transradial catheterization with a 7F sheath. Two-hundred patients, both men and women, will be recruited to the study.

Inclusion and exclusion criteria:

Two-hundred Hebrew-speaking subjects (male and female) who have previously undergone 7F transradial cardiac catheterization at the Lady Davis Carmel Medical Center between 1999 and 2012 will be contacted. Upon giving informed consent they will be recruited to the study.

Statistical analysis Univariate and multivariate analysis will be performed in order to identify demographic, clinical and procedural characteristics that are associated with radial artery occlusion.

References

1. Amoroso et al. Transradial access for primary percutaneous coronary intervention: the next standard of care? Heart 2010;96:1341-1344.
2. Freestone et al. Transradial cardiac procedures: The state of the art. Heart 2010;96:883-891.
3. Bertrand et al. Transradial Approach for Coronary Angiography and Interventions: Results of the First International Transradial Practice Survey. JACC Intv. 2010;3;1022-1031.
4. Pancholy et al. Effect of Duration of Hemostatic Compression on Radial Artery Occlusion After Transradial Access. CCI 2012;79:78-81.
5. Uhlemann et al. The Leipzig Prospective Vascular Ultrasound Registry in Radial Artery Catheterization. JACC Intv 2012;5:36-43.

ELIGIBILITY:
Inclusion Criteria:

* Previous transradial catheterization with a 7F vascular sheath

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two-hundred subjects who have previously undergone transradial cathetrization between the years 1999 and 2012 with a 7F sheath will be identified in the Lady Davis Carmel Medical Center Catheterization laboratory computerized database.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Normal reverse Allen test | Within 2 years of the initial procedure
  Radial artery patency will be studied with the reverse Allen test. This test is performed by simultaneously occluding both the radial and ulnar arteries until no pulse signal is detected with a pulse oximeter placed on the index finger. The pressure on the radial artery is then released and reappearance of the pulse signal on the oximeter is documented-signifying antegrade flow in the radial artery. This test is not associated with any reported complications or morbidity.

SECONDARY OUTCOMES:
Antegrade flow in the radial artery by ultrasound | Within 2 years of the initial procedure
  Radial artery flow will be studied with Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Jaffe, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Amoroso G, Kiemeneij F. Transradial access for primary percutaneous coronary intervention: the next standard of care? Heart. 2010 Sep;96(17):1341-4. doi: 10.1136/hrt.2010.196824. PMID 20801852
- [Background] Freestone B, Nolan J. Transradial cardiac procedures: the state of the art. Heart. 2010 Jun;96(11):883-91. doi: 10.1136/hrt.2007.134213. No abstract available. PMID 20478867
- [Background] Bertrand OF, Rao SV, Pancholy S, Jolly SS, Rodes-Cabau J, Larose E, Costerousse O, Hamon M, Mann T. Transradial approach for coronary angiography and interventions: results of the first international transradial practice survey. JACC Cardiovasc Interv. 2010 Oct;3(10):1022-31. doi: 10.1016/j.jcin.2010.07.013. PMID 20965460
- [Background] Pancholy SB, Patel TM. Effect of duration of hemostatic compression on radial artery occlusion after transradial access. Catheter Cardiovasc Interv. 2012 Jan 1;79(1):78-81. doi: 10.1002/ccd.22963. Epub 2011 May 16. PMID 21584923
- [Background] Uhlemann M, Mobius-Winkler S, Mende M, Eitel I, Fuernau G, Sandri M, Adams V, Thiele H, Linke A, Schuler G, Gielen S. The Leipzig prospective vascular ultrasound registry in radial artery catheterization: impact of sheath size on vascular complications. JACC Cardiovasc Interv. 2012 Jan;5(1):36-43. doi: 10.1016/j.jcin.2011.08.011. PMID 22230148